CLINICAL TRIAL: NCT05556135
Title: Role Of Serum Adiponectin In The Ealy Detection Of Renal Impairment In Patients With Non Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Abdelrafe Sayed, mohamed elyamany, Assiut University
Other Study IDs: Serum Adiponectin in NAFLD
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: NAFLD patients
  Interventions: Diagnostic Test: level of serun adiponectin
- group 2: non NAFLD patients
  Interventions: Diagnostic Test: level of serun adiponectin

INTERVENTIONS:
Diagnostic Test: level of serun adiponectin — estimation of level of serum adiponectin in NAFLD for early detection of renal impairement

SUMMARY:
Early detection of renal impairment in patients with Non-alcoholic fatty liver disease and its correlation with serum Adiponectin level.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) includes different types of liver damage, ranging from simple steatosis and nonalcoholic steatohepatitis (NASH) to liver cirrhosis and even hepatocellular carcinoma.(1) NAFLD is diagnosed by the presence of more than 5% fat accumulation in liver cells after excluding excessive alcohol intake in patients as well as other secondary causes of liver disease, such as drug-induced liver injury, viral and autoimmune hepatitis.(2) The diagnostic criteria for chronic kidney disease (CKD) are either the reduced estimated glomerular filtration rate (eGFR) (<60 mL/min/1.732) and/or abnormal albuminuria and/or overt proteinuria in patients for at least 3 months.(3) The association between NAFLD and CKD has recently attracted the attention of many experts. NAFLD and CKD share some common pathophysiological mechanisms as well as some metabolic risk factors for cardiovascular disease. Some studies have confirmed that the presence of NAFLD increases the risk of CKD and that the degree of liver fibrosis is related to CKD stage,(4) It is crucial to detect early renal impairment in patients with NAFLD to prevent CKD progression, minimize complications, and improve survival (1) Adiponectin is a recently identified adipose tissue-derived protein (adipocytokine) with important metabolic ,antiinflammatory, anti-atherogenic, and reactive oxygen species protective actions.(4) Adiponectin is one of the key regulators involved in glucose and lipid metabolism. Further analyses have shown its anti-inflammatory and anti-apoptotic roles in human cells.

Data from large cross sectional studies showed a positive correlation between serum Adiponectin and mortality in chronic kidney disease.(5)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with fatty liver aged from 18 to 60 yrs either diabetic or not .
2. Patient with normal echogenic kidney in ultrasound and eGFR more than 60 mL/min/1.73m2.
3. The Control group are completely healthy subjects without any systemic or liver and kidney affection

Exclusion Criteria:

* 1)Patients less than 18 yrs & more than 60 yrs 2)All patients having any other causes of renal and hepatic disease rather than Diabetes and having any other systemic problem.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All patients who fulfil inclusion and exclusion criteria then directed to nephrology unit to do other full investigations ,will be included in this study .
  1)Full history and clinical examination .2) Investigation :
  * All patients will be investigated for detection of renal impairment by :
    1)microalbuminurea.
    * 2)Urine analyses.
    * 3)Kidney function tests.
    * 4)calculate GFR.
    * 5)Complete blood count .
  * And also to detect the degree of liver affection by:
    * 1)liver function tests .
    * 2)abdominal ultrasound to grade fatty liver & determine echogenicity of kidney .
    * 3)Non-invasive blood test to detect degree of hepatic steatosis ( FIB-4 , APRI, fibrosis score ).
      4)fibroscane .
  * Detection of serum Adiponectin by ELISA technique using (EIA-3418) KIT, DRG international inc., USA *Investigations to control risk factors of Non-alcoholic fatty liver disease: -Calculate Body Mass Index (BMI). - Measuring the fasting blood sugar and HbA1C level in all subjects. -Lipid Profile.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Correlate serum Adiponectin level with renal impairment in non-alcoholic fatty liver disease. | baseline
  Correlate serum Adiponectin level with renal impairment in non-alcoholic fatty liver disease. /

CONTACTS AND LOCATIONS:
Overall Officials: mohamed hassan, MD, Study Director — master

REFERENCES:
- [Background] Montesano R, Orci L, Vassalli P. In vitro rapid organization of endothelial cells into capillary-like networks is promoted by collagen matrices. J Cell Biol. 1983 Nov;97(5 Pt 1):1648-52. doi: 10.1083/jcb.97.5.1648. PMID 6630296
- [Background] Stefan N, Stumvoll M. Adiponectin--its role in metabolism and beyond. Horm Metab Res. 2002 Sep;34(9):469-74. doi: 10.1055/s-2002-34785. PMID 12384822